CLINICAL TRIAL: NCT05390905
Title: A Multi-Center, Randomized, Double-Blind, Placebo/Active-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of HSK21542 Injection for Postoperative Pain Treatment
Brief Title: A Clinical Trial Evaluating the Efficacy and Safety of HSK21542 in Patients for Postoperative Pain Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK21542-303
Record Dates: First submitted 2022-05-12; First posted 2022-05-25 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK21542 (Experimental): HSK21542 injection
  Interventions: Drug: HSK21542 Injection
- tramadol (Experimental): Tramadol hydrochloride injection
  Interventions: Drug: Tramadol hydrochloride
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HSK21542 Injection — 1μg/kg/dose
  Other Names: HSK21542
  Arms: HSK21542
Drug: Tramadol hydrochloride — 50mg/dose
  Other Names: Tramadol
  Arms: tramadol
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo/active-controlled study. About 387 subjects undergoing elective abdominal operation under general anesthesia are planned to be enrolled and randomized into the HSK21542 group (129 subjects), tramadol group (129 subjects), and placebo group (129 subjects).

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤ age ≤ 70 years old, male or female;
2. The American Society of Anesthesiologists (ASA) Class I-II;
3. 18 kg/m2 ≤ BMI (body mass index) ≤ 40 kg/m2;
4. Subjects undergoing elective abdominal operation under general anesthesia (including laparoscopic surgery);
5. Subjects with an NRS score ≥ 4 at rest within 4 h after the surgery (when the last stitch of suture is completed) determined by investigators;
6. Subjects who agree to participate in this trial and voluntarily sign the informed consent form.

Exclusion Criteria:

Previous and concomitant diseases

1. Subjects with a history or evidence of any of the following diseases before screening:

1. History of cardiovascular diseases: uncontrolled hypertension (systolic blood pressure [SBP] ≥ 170 mmHg and/or diastolic blood pressure [DBP] ≥ 105 mmHg without treatment, or SBP > 160 mmHg and/or DBP > 100 mmHg despite antihypertensive treatment), aneurysm, serious arrhythmia, heart failure, Adams-stokes syndrome, the New York Heart Association (NYHA) Class ≥ III, serious superior vena cava syndrome, serious pericardial effusion, acute myocardial ischemia, unstable angina, myocardial infarction within 6 months before screening, history of tachycardia/bradycardia requiring medical treatment, II-III degree atrioventricular block (excluding subjects with pacemakers);
2. History of respiratory system disorders: serious chronic obstructive pulmonary disease, acute exacerbation of chronic obstructive pulmonary disease, serious airway stenosis, throat mass, history of tracheoesophageal fistula or airway tear, serious respiratory infection within 2 weeks before screening;
3. History of neurologic and psychiatric disorders: craniocerebral injury, convulsions, intracranial hypertension, cerebral aneurysms, history of cerebrovascular accidents; schizophrenia, mania, insanity, long-term use of psychotropic drugs, and history of cognitive dysfunction; history of depression, anxiety, and epilepsy, etc.;
4. History of acute poisoning with alcohol, hypnotics, analgesics, or other central nervous system acting drugs;
5. History of any major surgery within 3 months before screening, which may affect postoperative pain assessment as judged by investigators.

Past and concomitant medications 2. Known allergies or contraindications to opiates and other drugs that might be used in the clinical trial such as anesthetics (propofol/sevoflurane), muscle relaxants (cisatracurium), antiemetics (tropisetron); 3. Receipt of any one of the following medications or treatments at screening(with the exception of drugs specified in the protocol):

1. Use of opioid and non-opioid (such as paracetamol, aspirin [daily dose > 100 mg], indometacin, diclofenac, parecoxib sodium, and other non-steroidal anti-inflammatory drugs) analgesics with the interval between the last administration and randomization shorter than 5 half-lives of the drug or the duration of response (whichever is longer);
2. Consecutive use of opioid analgesics for any reason of more than 10 days within 3 months before screening;
3. Use of drugs with unknown half-lives that affect the analgesic effects within 14 days before randomization, or use of drugs that affect the analgesic effects with the interval between the last administration and randomization within 5 half-lives or duration of drug effect (calculated at maximum) (as per the packaging insert); such drugs include but are not limited to: sedative hypnotics (benzodiazepines [triazolam, diazepam, midazolam, etc.], non-benzodiazepines [zolpidem, zopiclone, zaleplon, etc.]), sedative anesthetics (anesthetic ether, nitrous oxide, sodium thiopental, ketamine, etomidate, etc.), glucocorticoids (dexamethasone hydrochloride, methylprednisolone, etc.), antiepileptics (carbamazepine, sodium valproate, etc.), anxiolytics (chlordiazepoxide, diazepam, etc.), antidepressants (imipramine, amitriptyline, etc.), and Chinese herbal medicines or Chinese patent medicines that may affect efficacy evaluation as judged by investigators;
4. Use of diuretics and compound drugs containing diuretics with the interval between the last administration and randomization shorter than 5 half-lives of the drug or the duration of response (whichever is longer).

Laboratory and other tests 4. The laboratory test parameters measured at screening reach one of the following criteria:

1. White blood cell count < 3.0 x 109/L;
2. Platelet count < 80 x 109/L;
3. Hemoglobin < 70 g/L;
4. Prolongation of prothrombin time (PT) exceeding the upper limit of normal (ULN) for 3 seconds;
5. Prolongation of activated partial thromboplastin time (APTT) exceeding the ULN for 10 seconds;
6. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2 x ULN;
7. Total bilirubin > 1.5 x ULN;
8. Blood creatinine > 1.5 x ULN;
9. Fasting blood glucose ≥ 11.1 mmol/L; 5. Positive for hepatitis C antibody (HCVAb), syphilis antibody, or human immunodeficiency virus (HIV) antibody at screening; Other circumstances 6. History of medication abuse, drug abuse, or alcohol abuse within 3 months before screening (alcohol abuse is defined as average daily alcohol drinking > 2 units of alcohol [1 unit = 360 mL of beer with 5% alcohol, 45 mL of liquor with 40% alcohol, or 150 mL of wine]); 7. History of blood donation or blood loss of ≥ 400 mL within 3 months before screening; 8. Participation in other clinical trials within 3 months before screening (defined as the receipt of investigational product or placebo); 9. Pregnant or breastfeeding females; females of child-bearing potential or males who are reluctant to use contraception during the trial; or subjects who are planning pregnancy within 3 months after the completion of the trial (including male subjects); 10. Subjects judged by investigators to have any other factors unsuitable for participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Sum of Pain Intensity Differences (SPID) in the HSK21542 group and the placebo group | From administration until 24 hours after administration
  Time-weighted SPID at rest within 0-24 h after the first administration in the HSK21542 group and the placebo group
Sum of Pain Intensity Differences (SPID) in tramadol group and the placebo group | From administration until 24 hours after administration
  Time-weighted SPID at rest within 0-24 h after the first administration in the tramadol group and the placebo group
Sum of Pain Intensity Differences (SPID) in the HSK21542 group and the tramadol group | From administration until 24 hours after administration
  Time-weighted SPID at rest within 0-24 h after the first administration in the HSK21542 group and the tramadol group

SECONDARY OUTCOMES:
Use of remedial analgesics within 0-12 h | From administration until 12 hours after administration
  Cumulative used amount of remedial analgesics within 0-12 h after the first administration, percentage of subjects not using remedial analgesics, and start time of remedial analgesic use
Use of remedial analgesics within 0-24 h | From administration until 24 hours after administration
  Cumulative used amount of remedial analgesics within 0-24 h after the first administration, percentage of subjects not using remedial analgesics, and start time of remedial analgesic use
Sum of Pain Intensity Differences (SPID) in each group | From administration until 12 hours after administration
  Time-weighted SPID at rest within 0-12 h after the first administration
Pain intensity difference (PID) | From administration until 24 hours after administration
  The PID at rest at each scoring time point after the first administration
Numerical rating scale（NRS）in each group | From administration until 24 hours after administration
  The NRS score at each scoring time point after the first administration
Numerical rating scale（NRS）at 0-12 h | From administration until 12 hours after administration
  The ratio of subjects with NRS score ≤ 3 for resting pain at 0-12 h after the first administration
Numerical rating scale（NRS）at 0-24 h | From administration until 24 hours after administration
  The ratio of subjects with NRS score ≤ 3 for resting pain at 0-24 h after the first administration
Duration of analgesia after the first administration | From administration until 24 hours after administration
  duration of NRS score ≤ 3 within 24 h after the first postoperative administration or the sum of the duration of NRS score ≤ 3 with fluctuations in pain within 24 h
Satisfaction scores on postoperative analgesia | From administration until 24 hours after administration
  Subject satisfaction score and investigator satisfaction score on postoperative analgesia at 24 h after the first administration

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong U, Wuhan, China

REFERENCES:
- [Derived] Zhong Y, Xu Y, Lei Q, Yang M, Wang S, Hu X, Xie H, Li Y, Qin Z, Gu Z, Zhang J, Wang Y, Wu J, Wang H, Ming Y, Xia Z, Zhai H, Jiang K, Zhang P, Wang Z, Wang L, Li L, Cheng Z, Jiang H, Wang G, Chen J, Zhao Z, Chen X, Yan M. HSK21542 in patients with postoperative pain: two phase 3, multicentre, double-blind, randomized, controlled trials. Nat Commun. 2025 May 24;16(1):4830. doi: 10.1038/s41467-025-60013-y. PMID 40413233